CLINICAL TRIAL: NCT00160680
Title: A Pilot, Open, Monocenter, Randomized Two Parallel Groups, Clinical Efficacy Trial: Comparison Continuous Versus on Demand Regimen of Treatment With Levocetirizine 5 mg Oral Tablets, Once a Day, in Adults Suffering From Persistent Allergic Rhinitis (PER) Over 6 Months
Brief Title: ATAREAL (Antihistamine Treatment for Allergic Rhinitis in Real Life)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB S.A. - Pharma Sector (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A00392; 2004-003858-26 (EudraCT Number)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Persistent Allergic Rhinitis; HDM; Parietaria; sneezing; rhinorrhea; ocular pruritus; Rhinasthma; inflammatory cells; ICAM-1; ATAREAL; Xyzal; Levocetirizine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Sneezing; Rhinorrhea | interventions — levocetirizine

ARMS (2):
- Continuous Treatment (Experimental): 5 mg of Levocetirizine (LCTZ) was taken orally once a day.
  Interventions: Drug: Levocetirizine
- On Demand Treatment (Experimental): 5 mg of Levocetirizine (LCTZ) was taken whenever needed.
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — * Pharmaceutical form: Tablet
  * Concentration: 5 mg
  * Route of administration: Oral use
  Other Names: Xyzal

SUMMARY:
Comparison of clinical efficacy and safety of levocetirizine in PER continuous versus on demand, measured by evolution of individual symptom scores during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of Persistent allergic Rhinitis (PER) requiring treatment known at least since 2 years.
* Positive skin prick test (wheal > 3 mm larger than the diluent control) or Radio Allergo Sorbent Assay (RAST) (>= 3.5 IU/ml) to House Dust Mite (HDM) and Parietaria (less than 1 year).
* Minimum mean Total 4 Symptom Score (T4SS) of 6 over baseline period.

Exclusion Criteria:

* Subjects currently treated by specific parietaria pollen immunotherapy
* Subjects suffering from non-allergic asthma
* Chronic use of inhaled steroids and/or long acting β2 agonists; and/or corticosteroids dependent asthma (severe asthma)
* Atopic dermatitis or urticaria requiring antihistamine treatment or the administration of oral or topical corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2006-06-01 (Actual); Study Completion 2006-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Genova, Italy

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in March 2005 and concluded in June 2006.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Continuous Treatment (CT): 5 mg of Levocetirizine (LCTZ) was taken orally once a day.
- On Demand Treatment (ODT): 5 mg of Levocetirizine (LCTZ) was taken whenever needed.
Period: Overall Study
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Started | 31 | 31
Completed | 22 | 18
Not Completed | 9 | 13
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 4 | 9

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat Population.
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT) | Total Title
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.74 (12.33) | 35.20 (10.71) | 34.97 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Total 4 Symptom Score (T4SS) During the Treatment Period
Description: The T4SS is the sum of the symptom scores for sneezing, rhinorrhea, nasal pruritus and ocular pruritus. Each of the symptoms is rated retrospectively over the past 24 hours using a 4-point 0 to 3 scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe). Total T4SS is the sum of the idividual scores and ranges from 0-12. Increasing values are associated with increasing severity of disease.
Time Frame: During the treatment period until week 24
Population: Only patients with a valid mean weekly T4SS during the treatment period were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 29 | 29
units on a scale | 2.89 (0.43) | 3.15 (0.44)
Statistical Analysis 1: Comparison: Continuous Treatment (CT) vs On Demand Treatment (ODT); Test type: Superiority or Other; p = 0.667, ANCOVA; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.96 to 1.50]

2. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 1 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 1 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 1 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 28 | 29
units on a scale | 4.55 (0.61) | 3.83 (0.61)

3. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 2 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 2 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 2 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 27 | 26
units on a scale | 4.04 (0.63) | 3.14 (0.63)

4. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 3 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 3 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 3 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 25 | 24
units on a scale | 2.98 (0.50) | 2.58 (0.51)

5. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 4 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 4 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 4 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 26 | 20
units on a scale | 2.47 (0.47) | 2.67 (0.50)

6. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 5 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 5 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 5 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 22 | 18
units on a scale | 1.74 (0.45) | 3.31 (0.48)

7. Secondary Outcome: Mean Monthly Total 4 Symptom Score (T4SS) for Month 6 of the Treatment Period
Description: as for outcome 1
Time Frame: During month 6 of the 6 months treatment period
Population: Only patients with a valid T4SS at month 6 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 19 | 19
units on a scale | 2.19 (0.57) | 3.64 (0.59)

8. Secondary Outcome: Mean Weekly Individual Symptoms Scores During the Treatment Period
Description: Individual symptom scores include scores for Sneezing, Rhinorrhea, Nasal Pruritus, Ocular Pruritus, and Nasal Congestion.
  The subjects had to evaluate the severity of the symptoms retrospectively over the past 24 hours (0 = absent, 1 = mild, 2 = moderate, 3 = severe). Increasing scores are associated with increasing severity.
Time Frame: During the treatment period until week 24
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean weekly individual symptoms scores were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 30 | 30
  Sneezing Score | 0.82 (0.11) | 0.94 (0.12)
  Rhinorrhea Score: number analyzed (Participants) | 30 | 30
  Rhinorrhea Score | 0.80 (0.12) | 0.80 (0.12)
  Nasal Pruritus Score: number analyzed (Participants) | 29 | 30
  Nasal Pruritus Score | 0.71 (0.12) | 0.74 (0.12)
  Ocular Pruritus Score: number analyzed (Participants) | 29 | 29
  Ocular Pruritus Score | 0.55 (0.10) | 0.68 (0.10)
  Nasal Congestion Score: number analyzed (Participants) | 26 | 28
  Nasal Congestion Score | 0.87 (0.14) | 1.08 (0.14)

9. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 1 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 1 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 1 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 29 | 30
  Sneezing Score | 1.31 (0.15) | 1.12 (0.15)
  Rhinorrhea Score: number analyzed (Participants) | 29 | 30
  Rhinorrhea Score | 1.33 (0.16) | 0.93 (0.16)
  Nasal Pruritus Score: number analyzed (Participants) | 28 | 30
  Nasal Pruritus Score | 1.06 (0.17) | 0.97 (0.16)
  Ocular Pruritus Score: number analyzed (Participants) | 28 | 29
  Ocular Pruritus Score | 0.90 (0.17) | 0.86 (0.17)
  Nasal Congestion Score: number analyzed (Participants) | 24 | 28
  Nasal Congestion Score | 1.25 (0.19) | 1.25 (0.18)

10. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 2 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 2 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 2 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 27 | 27
  Sneezing Score | 1.20 (0.16) | 0.87 (0.16)
  Rhinorrhea Score: number analyzed (Participants) | 27 | 26
  Rhinorrhea Score | 1.14 (0.17) | 0.80 (0.17)
  Nasal Pruritus Score: number analyzed (Participants) | 27 | 26
  Nasal Pruritus Score | 0.98 (0.16) | 0.75 (0.16)
  Ocular Pruritus Score: number analyzed (Participants) | 27 | 26
  Ocular Pruritus Score | 0.77 (0.17) | 0.77 (0.17)
  Nasal Congestion Score: number analyzed (Participants) | 24 | 25
  Nasal Congestion Score | 1.03 (0.19) | 1.04 (0.18)

11. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 3 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 3 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 3 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 25 | 24
  Sneezing Score | 0.82 (0.14) | 0.81 (0.15)
  Rhinorrhea Score: number analyzed (Participants) | 25 | 24
  Rhinorrhea Score | 0.84 (0.14) | 0.66 (0.14)
  Nasal Pruritus Score: number analyzed (Participants) | 25 | 24
  Nasal Pruritus Score | 0.74 (0.13) | 0.53 (0.13)
  Ocular Pruritus Score: number analyzed (Participants) | 25 | 24
  Ocular Pruritus Score | 0.61 (0.13) | 0.60 (0.14)
  Nasal Congestion Score: number analyzed (Participants) | 24 | 23
  Nasal Congestion Score | 0.87 (0.16) | 0.91 (0.16)

12. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 4 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 4 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 4 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 26 | 20
  Sneezing Score | 0.78 (0.14) | 0.85 (0.15)
  Rhinorrhea Score: number analyzed (Participants) | 26 | 20
  Rhinorrhea Score | 0.69 (0.14) | 0.72 (0.14)
  Nasal Pruritus Score: number analyzed (Participants) | 26 | 20
  Nasal Pruritus Score | 0.60 (0.13) | 0.59 (0.14)
  Ocular Pruritus Score: number analyzed (Participants) | 26 | 20
  Ocular Pruritus Score | 0.44 (0.11) | 0.53 (0.12)
  Nasal Congestion Score: number analyzed (Participants) | 25 | 19
  Nasal Congestion Score | 0.75 (0.15) | 1.07 (0.16)

13. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 5 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 5 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 5 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 22 | 18
  Sneezing Score | 0.51 (0.12) | 1.00 (0.13)
  Rhinorrhea Score: number analyzed (Participants) | 22 | 18
  Rhinorrhea Score | 0.51 (0.14) | 0.93 (0.15)
  Nasal Pruritus Score: number analyzed (Participants) | 22 | 18
  Nasal Pruritus Score | 0.44 (0.12) | 0.77 (0.13)
  Ocular Pruritus Score: number analyzed (Participants) | 22 | 18
  Ocular Pruritus Score | 0.27 (0.10) | 0.63 (0.11)
  Nasal Congestion Score: number analyzed (Participants) | 21 | 17
  Nasal Congestion Score | 0.63 (0.15) | 1.08 (0.16)

14. Secondary Outcome: Mean Monthly Individual Symptoms Scores During Month 6 of the Treatment Period
Description: as for outcome 8
Time Frame: During month 6 of the 6 months treatment period
Population: 31 patients were included in the ITT-Set for each treatment group. Only patients with valid mean monthly individual symptoms scores at month 6 were included in the analysis of this outcome measure. Number of patients analyzed are given for each individual symptoms score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Continuous Treatment (CT) | On Demand Treatment (ODT)
Number analyzed (Participants) | 31 | 31
units on a scale
  Sneezing Score: number analyzed (Participants) | 19 | 19
  Sneezing Score | 0.61 (0.15) | 1.11 (0.16)
  Rhinorrhea Score: number analyzed (Participants) | 19 | 19
  Rhinorrhea Score | 0.57 (0.15) | 1.00 (0.16)
  Nasal Pruritus Score: number analyzed (Participants) | 19 | 19
  Nasal Pruritus Score | 0.59 (0.15) | 0.84 (0.16)
  Ocular Pruritus Score: number analyzed (Participants) | 19 | 19
  Ocular Pruritus Score | 0.36 (0.14) | 0.69 (0.14)
  Nasal Congestion Score: number analyzed (Participants) | 18 | 18
  Nasal Congestion Score | 0.82 (0.17) | 1.15 (0.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 2 (Week 0) until Visit 9 (Week 24).
Description: Adverse Events refer to the Safety Population consisting of all randomized subjects. One subject took the treatment under on demand regimen instead of continuous regimen. For the safety analyses, this subject was analyzed according to actual regimen received. Therefore, the Safety Population consisted of 62 subjects: 30 under the continuous regimen and 32 under the on demand regimen.
Groups:
- Continuous Treatment (SS): 5 mg of Levocetirizine (LCTZ) was taken orally once a day.
- On Demand Treatment (SS): 5 mg of Levocetirizine (LCTZ) was taken whenever needed.
Arm/Group | Continuous Treatment (SS) | On Demand Treatment (SS)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 4/30 | 10/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Treatment (SS) (N=30) | On Demand Treatment (SS) (N=32)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days